CLINICAL TRIAL: NCT07231640
Title: PrOTECT AL: PrEP Optimization Through Enhanced Continuum Tracking
Acronym: PrOTECT AL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael J Mugavero, MD, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-300014665; R01MH136851-01A1 (NIH)
Record Dates: First submitted 2025-11-04; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: HIV; PrEP; PrEP Uptake; HIV Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrOTECT AL Implementation Strategy (Other): The PrOTECT AL dashboard consisted of a public-facing homepage with information on the purpose of the project, resources for finding PrEP services across the state, information on project partners, and reading materials on HIV and prevention efforts across AL. From the website, partners can access the data dashboard via a clinic-specific login where they view both aggregate data and their clinic-level data. Data elements include: number of patients referred for, linked to, prescribed, or discontinued from PrEP within the reporting period (3-month timeframe); primary PrEP indications recorded; and AL counties served. These elements can be filtered down by race, age, and gender. Additional proposed modifications, will include an PrEP coverage map, showing where the greatest unmet needs are for PrEP service delivery in the state as well as a PrEP equity scores, clinic performance indicator that will be populate every 3-months.
  Interventions: Other: PrOTECT AL Implementation Strategy

INTERVENTIONS:
Other: PrOTECT AL Implementation Strategy — with information on the purpose of the project, resources for finding PrEP services across the state, information on project partners, and reading materials on HIV and prevention efforts across AL. From the website, partners can access the data dashboard via a clinic-specific login where they view both aggregate data and their clinic-level data. Data elements include: number of patients referred for, linked to, prescribed, or discontinued from PrEP within the reporting period (3-month timeframe); primary PrEP indications recorded; and AL counties served. These elements can be filtered down by race, age, and gender. Additional proposed modifications, will include an PrEP coverage map, showing where the greatest unmet needs are for PrEP service delivery in the state as well as a PrEP equity scores, clinic performance indicator that will be populate every 3-months.

SUMMARY:
The purpose of this study is to enhance and evaluate the implementation of a PrEP Care Continuum data dashboard across seven distinct clinical sites in Alabama. By leveraging real-time data and fostering collaborative partnerships, this project aims to accurately visualize care disparities, allocate resources strategically, identify and address care gaps in the delivery of PrEP services, and gauge its impact on HIV prevention efforts.

DETAILED DESCRIPTION:
Aim 1: Conduct data mapping procedures to inform real-time data capture at agencies providing PrEP (n = 7) and refine the PrOTECT AL dashboard with practice transformation implementation strategies.

Sub-aim 1a: Refine the dashboard through incorporation of 1) quarterly STI incidence data from ADPH overlapped with clinic-PrEP prescription data to aid in visualization of clinic service area PrEP coverage and 2) clinic PrEP equity performance indexes.

Sub-aim 1b: Conduct on-site assessment of organizational readiness via electronic surveys and checklists.

Aim 2: Evaluate implementation outcomes associated with deployment of the PrOTECT AL dashboard and practice transformation implementation strategies, grounded in RE-AIM. Implementation outcomes (e.g., reach, maintenance) will be evaluated at each site, with the primary implementation outcome being change over time of the proportion of PrEP prescriptions to Black persons with a PrEP indication (i.e., adoption based on PrEP coverage) relative to the proportion of PrEP prescriptions to White persons with a PrEP indication.

Aim 3: Evaluate the effectiveness of PrOTECT AL by conducting an interrupted, time-series study of PrEP-to-need ratio (PNR) and PrEP coverage. Investigators will evaluate the hypothesis that implementation of the PrOTECT AL dashboard will result in greater than expected increase in PNR and PrEP coverage.

ELIGIBILITY:
Inclusion Criteria:

* currently practicing providers (either a clinician, nurse or medical assistant), OR 2) clinical administrator (e.g., someone in a leadership role within the PrEP clinic), OR 3) a data manager (i.e., someone who collects, enters and or manages data within the clinic) AND
* English speaking
* Age ≥ 18.

Exclusion Criteria:

* Not one of the seven participating sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Adoption | Quarterly from baseline to 36 months
  The primary outcome is the change over time of the proportion of PrEP prescriptions to Black persons with a PrEP indication (i.e. PrEP coverage) compared to the proportion of PrEP prescriptions to White persons with a PrEP indication.

SECONDARY OUTCOMES:
Public Health Impact | Baseline, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months post-baseline
  Investigators will conduct segmented linear regression models to compare PrEP-to-need ration (PNR) and PrEP coverage in AL in the pre and post dashboard intervention phases, with PNR and PrEP coverage assessed in 6-month intervals.

OTHER OUTCOMES:
Reach | Quarterly from baseline to 36 months
  The number of PrEP prescriptions at the clinic-level and evaluating if there is increase in prescriptions over time.
Acceptability of the intervention | Baseline, 18-months, 36- months
  Investigators will conduct internet-based surveys to assess clinic member attitudes regarding the acceptability of prescribing PrEP and the dashboard. Survey measures are based on a validated survey instrument, the Acceptability of Intervention Measure (AIM)
Maintenance | 36 months
  Using the administrative web-metric data, investigators will examine longitudinal patterns in dashboard use for each clinic to determine whether changes in behaviors were sustained over time, using the Clinical Sustainability Assessment Tool (CSAT)
Feasibility of the intervention | baseline, 18-months, 36-months
  Investigators will conduct internet-based surveys to assess clinic member attitudes regarding the feasibility of prescribing PrEP and the dashboard. Survey measures are based on a validated survey instrument, the Feasibility of Intervention Measure (FIM).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mugavero, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No